CLINICAL TRIAL: NCT02591563
Title: A Study Evaluating Pathogens and Immunity to Acute Otitis Media and Nasopharyngeal Colonization in Healthy Children.
Brief Title: Evaluate Pathogens and Immunity to Acute Otitis Media in Healthy Children.
Acronym: AOM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Rochester General Hospital (Other)
Responsible Party: Principal Investigator, Michael Pichichero, MD, Director, Rochester General Hospital Research Institute, Rochester General Hospital
Other Study IDs: CIC 1141 B-09-1
Record Dates: First submitted 2015-10-28; First posted 2015-10-29 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Nasopharyngeal Colonization and Acute Otitis Media
MeSH Terms: conditions — Otitis Media | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — middle ear fluid, nasal swabs, nasal wash, and blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Healthy children: 6-36 months of age who will have the following study procedures: Venipuncture, Nasopharyngeal swab, nasopharyngeal wash, tympanocentesis
  Interventions: Other: procedures

INTERVENTIONS:
Other: procedures — Nasopharyngeal swab, nasopharyngeal wash, tympanocentesis (if acute otitis media occurs), venipuncture

SUMMARY:
The purpose of this study is to Evaluate Pathogens and Immunity to Acute Otitis Media in Healthy Children.

DETAILED DESCRIPTION:
A prospective evaluation of bacterial pathogens Streptococcus. pneumoniae, Haemophilus influenzae, Moraxella. catarrhalis and Staphylococcus aureus and their antibiotic susceptibility when colonizing the nasopharynx and/or causing acute otitis media in the years 2015-2025. The goal will be to recruit children into a prospective group beginning at 6 months of age and followed to 36 months of age in suburban Rochester, New York. Nasopharyngeal and nasal wash samples will be obtained at each well child visit and at acute otitis media (AOM) episodes. Middle ear fluid will be obtained from every child with an acute otitis media episode who undergoes a tympanocentesis procedure. All of the nasopharyngeal and middle ear fluid samples collected will be tested by standard microbiologic techniques to identify the presence of 4 potential otopathogens (S. pneumoniae, H. influenzae, M. catarrhalis and S. aureus). All S. pneumoniae will undergo serotyping and antibiotic susceptibility testing. All samples that are culture negative will be evaluated with a multi-locus PCR test to examine for presence of potential otopathogens.

ELIGIBILITY:
Inclusion Criteria:

Healthy Children:

* Male or female age greater than/equal to 6 months or less than/equal to 36 months old.
* Parent/guardian willing to bring to all study visits

Exclusion Criteria:

* Any major illness/condition that in investigator opinion would put subject at risk during study.
* Otorrhea or tympanostomy tubes present in either ear @ time of enrollment.
* Direct descendant of study site personnel.
* Subjects < 6 months old or >36 months old at the time of enrollment

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy 6-36 month old children or Acute Otitis Media diagnosed children >/= 6mo but </= 36 months
Sampling Method: Non-Probability Sample
Enrollment: 1320 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The distribution of bacteria causing acute otitis media. | 10 years
  In this study, we are exploring the three main bacteria (Streptococcus pneumoniae, Haemophilus influenzae, Moraxella catarrhalis) isolated from middle ear fluid samples (obtained by tympanocentesis) during acute otitis media episode in children ages 6-36 months.

SECONDARY OUTCOMES:
The distribution of potential otopathogens colonizing the nasopharynx. | 10 years
  In this study we are exploring the three main bacteria (Streptococcus pneumoniae, Haemophilus influenzae, Moraxella catarrhalis) isolated from nasopharynx of children during their routine healthy visits at 6-36 months of age during an AOM episode.

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Pichichero, MD, Principal Investigator — Rochester General Hospital
Locations (1):
- Rochester General Hospital, Rochester, New York, United States